CLINICAL TRIAL: NCT02340039
Title: The Acute Effects of Blackcurrant and Apple Extracts on Postprandial Glycaemia: a Randomised Controlled Trial. The GLU-FRU Study
Brief Title: Effects of Fruit Extracts on Glycaemia: The GLU-FRU Study
Acronym: GLU-FRU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Principal Investigator, Dr Wendy Hall, Lecturer in Nutritional Sciences, King's College London
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GF2015
Record Dates: First submitted 2015-01-13; First posted 2015-01-16 (Estimated); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Postprandial Hyperglycemia
Keywords: Polyphenol; Fruit; Metabolic
MeSH Terms: conditions — Hyperglycemia | interventions — Polyphenols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Blackcurrant &Apple (Experimental): 600 mg blackcurrant anthocyanins + 600 mg apple polyphenols delivered in a low sugar fruit drink
  Interventions: Dietary Supplement: Polyphenols
- Apple (Experimental): 1200 mg apple polyphenols delivered in a low sugar fruit drink
  Interventions: Dietary Supplement: Polyphenols
- Control drink (Placebo Comparator): No polyphenols delivered in a low sugar fruit drink
  Interventions: Dietary Supplement: Polyphenols

INTERVENTIONS:
Dietary Supplement: Polyphenols — Drinks will be delivered in random order at 3 separate study visits immediately before a high-carbohydrate meal. Seven days wash-out period will be required between study days.

SUMMARY:
Raised blood glucose levels can lead to adverse modifications to functional proteins within the body and eventually lead to the development of type 2 diabetes. Fruit polyphenols may help to control glycaemia following a carbohydrate meal or beverage. The aim of this study is to investigate the effects of blackcurrant (BC) and apple (A) extracts on postprandial glycaemia, insulinaemia and plasma gastric inhibitory polypeptide concentrations following a mixed carbohydrate test meal.

DETAILED DESCRIPTION:
Introduction:

Diets with a high glycaemic load (a measure of the overall blood glucose-raising effect of a serving of a food) and containing high amounts of non-milk extrinsic sugars may contribute towards increased risk of developing type 2 diabetes (T2D). Raised blood glucose levels can lead to adverse modifications to functional proteins within the body and eventually lead to the development of T2D. Large peaks in blood glucose after a meal are a risk factor for T2D, and therefore it is desirable to consume a diet that will allow more gradual rises in blood glucose levels after meals. Fruit polyphenols may help to control glycaemia following a carbohydrate meal or beverage. Possible mechanisms include inhibition of intestinal enzymes and inhibition of intestinal glucose absorption by decreasing SGLT1/GLUT2 transport activity. The scientific literature also suggests that foods rich in polyphenols exert beneficial effects on risk factors of cardiovascular disease such as hypertension, lipid metabolism and vascular function.

Study Design:

A randomised, controlled, double-blind, cross-over study will be conducted. Subjects will receive combined blackcurrant and apple polyphenols, apple polyphenols only or placebo in random order at 3 separate study visits immediately before a high-carbohydrate meal. Seven days wash-out period will be required between study days.Standardised diet and exercise advice will be given prior to the visit. Subjects will arrive on each study visit between 09.00 and 10.00 h, after a 12 h overnight fast. They will then be cannulated in a forearm vein and baseline fasting blood samples will be taken in duplicate. All test drinks will be blended to be equal in volume, macronutrient and energy content. Fruit extracts instead of whole fruits will be administered to avoid the confounding effect of fruit fibre/viscosity on gastric emptying rate. Following consumption of the test drink, the high carbohydrate meal (starch and sucrose) will be served (white bread with apricot jam). Outcome variables will be measured postprandially until 120 min post-meal.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-60 y
* Male and female (post-menopausal only)
* Healthy (free of diagnosed diseases in the exclusion criteria)
* BMI 18-35 kg/m2
* Able to understand the information sheet and willing to comply with study protocol
* Able to give informed written consent

Exclusion Criteria:

* Those diagnosed with Phenylketonuria (PKU),
* Those with known or suspected food intolerances, allergies or hypersensitivity
* Women who are known to be pregnant or who are intending to become pregnant over the course of the study
* Women who are breast feeding
* Participation in another clinical trial
* Those who have donated blood within 3 months of the screening visit and participants for whom participation in this study would result in having donated more than 1500 millilitres of blood in the previous 12 months.
* Those with Full Blood Counts and Liver Function test results outside of the normal range (see table 1 below).
* Pre-menopausal women due to the potential influence of cyclical changes in reproductive hormones on insulin sensitivity
* Current smokers, or reported giving up smoking within the last 6 months
* History of substance abuse or alcoholism
* Reported history of CVD, diabetes (or fasting glucose ≥ 7.1 mmol/L), cancer, kidney, liver or bowel disease, gastrointestinal disorder or use of drug likely to alter gastrointestinal function
* Unwilling to restrict consumption of specified high polyphenol foods for 24 h before the study
* Weight loss >3kg in preceding 2 months and body mass index <18 or >35 kg/m2
* Blood pressure ≥160/100 mmHg
* Total cholesterol ≥ 7.5 mmol/L; fasting triacylglycerol concentrations ≥ 5.0 mmol/L
* Medications that may interfere with the study such as alpha-glucosidase inhibitors (acarbose: Glucobay), insulin-sensitising drugs (metformin: Glucophage, Glucophage SR, Eucreas, Janumet; thiazolidinediones: Actos, Competact), sulfonylureas (Daonil, Diamicron MR, Glibenese, Minodiab, Amaryl Tolbutamide), and lipid-lowering drugs (statins, nicotinic acid, colestyramine anhydrous, ezetimibe, fibrates). Other medications should be reviewed by medical representative from KCL on a case by case basis.
* Nutritional supplements that may interfere with the study such as higher dose vitamins/minerals (>200% RNI), B vitamins, Vitamin C, calcium, copper, chromium, iodine, iron, magnesium, manganese, phosphorus, potassium and zinc. Subjects already taking vitamin or minerals at a dose around 100% or less up to 200% of the RNI, or evening primrose/algal/fish oil supplements will be asked to maintain habitual intake patterns, ensuring that they take them every day and not sporadically. They will be advised not to stop taking supplements or start taking new supplements during the course of the study.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2015-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Postprandial glycaemia | baseline and 10, 20, 30, 45, 60, 75, 90 and 120 min following the test drink.
  Peak postprandial plasma glucose concentrations (Cmax) t +0-30 min and change from baseline data and areas over baseline t+0-30 min and t+0-120 min

SECONDARY OUTCOMES:
Postprandial insulinaemia | baseline and 10, 20, 30, 45, 60, 75, 90 and 120 min following the test drink.
  Peak postprandial insulin concentrations (Cmax) t +0-30 min and change from baseline data and areas over baseline t+0-30 min and t+0-120 min
Postprandial glucose-dependent insulinotropic polypeptide (GIP) concentrations | baseline and 10, 20, 30, 45, 60, 75, 90 and 120 min following the test drink.
  Peak postprandial GIP concentrations (Cmax) t +0-30 min and change from baseline data and areas over baseline t+0-30 min and t+0-120 min
Postprandial glucagon-like peptide-1 (GLP-1) concentrations | baseline and 10, 20, 30, 45, 60, 75, 90 and 120 min following the test drink.
  Peak postprandial GLP-1 concentrations (Cmax) t +0-30 min and change from baseline data and areas over baseline t+0-30 min and t+0-120 min
Blood pressure | baseline and 60, 90 and 120 min following the test drink.
  Change in the blood pressure after consumption of test drink
Vascular function (Digital Volume Pulse; DVP) | baseline and 60, 90 and 120 min following the test drink.
  Change in the tone of larger arteries (stiffness index) and small to medium-sized arteries (reflection index).
Plasma non-esterified fatty acids (NEFA) | baseline and 10, 20, 30, 45, 60, 75, 90 and 120 min following the test drink.
  Peak postprandial NEFA concentrations (Cmax) t +0-30 min and change from baseline data and areas over baseline t+0-30 min and t+0-120 min
Plasma triglycerides (TAG) | baseline and 10, 20, 30, 45, 60, 75, 90 and 120 min following the test drink.
  Peak postprandial TAG concentrations (Cmax) t +0-30 min and change from baseline data and areas over baseline t+0-30 min and t+0-120 min

CONTACTS AND LOCATIONS:
Overall Officials: Wendy L Hall, Dr, Principal Investigator — King's College London
Locations (1):
- Metabolic Research Unit at King's College London. Franklin-Wilkins Buiding. Waterloo Campus, London, England, United Kingdom

REFERENCES:
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/28886437